CLINICAL TRIAL: NCT06092970
Title: Clinical Protocol REN-007E - Extension Study: An Evaluation of Patient Reported Outcomes and Clinical Outcomes Through 12 Months Post-Cardiac Surgery in Subjects Enrolled in Study REN-007
Brief Title: An Evaluation of Patient Reported Outcomes and Clinical Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REN-007E
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Post-Operative Complications in Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RBT-1: Patients undergoing CABG, valve, or combined CABG/valve surgery
  Interventions: Drug: RBT-1
- Placebo: Patients undergoing CABG, valve, or combined CABG/valve surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBT-1 — Intravenous administration
  Groups: RBT-1
Drug: Placebo — Intravenous administration
  Groups: Placebo

SUMMARY:
This extension study is being conducted to assess the following objectives through 12 months post-cardiac surgery:

* Patient reported outcomes (PRO), using the EQ-5D questionnaire
* Clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed the REN-007 study to be eligible to participate in the Extension Study.

Exclusion Criteria:

* Subjects who did not complete the REN-007 study are not eligible to participate in the Extension Study.
* Female subjects who become pregnant during the REN-007 study are not eligible to participate in the Extension Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who complete the Phase 3 REN-007 study are eligible to participate in the Extension Study.
Sampling Method: Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation | 12 Months Post-Cardiac Surgery
  To evaluate patient reported outcomes (PRO) using the EQ-5D questionnaire
Evaluation | 12 Months Post-Cardiac Surgery
  The number of subjects with the following clinical outcomes will be reported
  Clinical Outcomes:
  * Chronic kidney disease (CKD) - new diagnosis
  * Acute kidney injury (AKI) or CKD requiring dialysis
  * Atrial fibrillation - new-onset
  * Death
  * Myocardial infarction (MI)
  * Non-fatal cardiac arrest
  * Readmission to hospital
  * Reoperation for coronary artery bypass graft (CABG) and/or valve dysfunction
  * Stroke

CONTACTS AND LOCATIONS:
Locations (35):
- United States (28):
  - Research Site, Huntsville, Alabama
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlantis, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - New York Presbyterian-Queens, Flushing, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
- Canada (7):
  - Research Site, Kelowna, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No